CLINICAL TRIAL: NCT03769207
Title: Evaluation of the Use of Apple Watch Features for Identification of Cardiac Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apple Inc. (Industry)
Responsible Party: Principal Investigator, Marco Perez, Assistant Professor of Medicine (Cardiovascular Medicine), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1.2; 48787 (Other: Stanford IRB)
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Atrial Flutter | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ambulatory ECG (Other)
  Interventions: Device: Ambulatory ECG

INTERVENTIONS:
Device: Ambulatory ECG — Eligible participants are asked to wear the ambulatory ECG monitor

SUMMARY:
This post-marketing study is conducted to characterize the ability of Apple Watch rhythm analysis software to identify Atrial Fibrillation (AF) and facilitate subsequent clinical evaluation among users who contact AppleCare.

ELIGIBILITY:
Inclusion Criteria:

1. Possession of the following at time of eligibility screening:

   * iPhone (5s or later) with iOS version 12.1.1 or later defined as iPhone model/iOS version used to complete screening eligibility.
   * Apple Watch (Series 1-4) with watchOS version 5.1.2 or later defined as Apple Watch model/watchOS paired with iPhone used to complete screening eligibility
2. At least one of the following by self-report before consent:

   * Irregular Rhythm Notification
   * ECG app classification of Atrial Fibrillation
   * ECG app classification of Inconclusive defined as "Inconclusive," "Heart Rate Over 120," or "Heart Rate Under 50"
3. Age ≥ 22 years at time of eligibility screening
4. Current resident of the United States at time of eligibility screening, and will reside in the United States for the length of the study
5. Proficient in written and spoken English
6. Valid phone number associated with iPhone, ascertained from self-report
7. Valid email address, ascertained from self-report

Exclusion Criteria:

1. Shared iCloud account
2. Shared AppleWatch

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco V Perez, MD, Principal Investigator — Stanford University; Minang (Mintu) Turakhia, MD, MAS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received an irregular pulse notification or who had an AF classification on the ECG app and then called the sponsor's customer support were invited to download the study app and enroll. They had a remote study visit, were sent an ECG patch to wear and return for analysis, and had a second remote visit to review the findings.
Period: Overall Study
Arm/Group | Ambulatory ECG
Started | 17
Attended First Study Visit | 11
ECG Patch Shipped | 11
ECG Patch Returned and Readable | 9
Attended Second Study Visit | 6
Completed | 6
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Ambulatory ECG
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  Asian | 1
  Middle Eeastern or North African | 1
  Preferred not to respond | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation or Atrial Flutter (AF) of at Least 30 Seconds Duration
Description: Detected on ambulatory ECG patch monitor for a participant who received an IRN or Apple Watch ECG app - AFib classification
Time Frame: During ambulatory ECG Monitoring (up to 8 days)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Ambulatory ECG
Number analyzed (Participants) | 9
Proportion of participants | 0.11 [0.003 to 0.48]

2. Secondary Outcome: Arrhythmias Other Than AF
Description: Detected on an ambulatory ECG patch monitor for a participant who received an IRN or Apple Watch ECG app - AFib classification
Time Frame: During ambulatory ECG Monitoring (up to 8 days)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Ambulatory ECG
Number analyzed (Participants) | 9
Proportion of participants | 0 [0 to 0]

3. Secondary Outcome: Self-reported Contact With Healthcare Provider
Time Frame: Between 15 to 90 days following enrollment
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Ambulatory ECG
Number analyzed (Participants) | 9
Proportion of participants | 0.56 [0.21 to 0.86]

ADVERSE EVENTS:
Time Frame: 9 months (participants may have reported adverse events at any time from enrollment to close of study)
Arm/Group | Ambulatory ECG
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambulatory ECG (N=17)
Anxiety (Psychiatric disorders) | 2 (2)
Elevated Heart Rate (Cardiac disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The small number of enrolled participants prevents us from drawing meaningful conclusions from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03769207/Prot_SAP_000.pdf